CLINICAL TRIAL: NCT04578067
Title: Økt Fysisk Aktivitet og Sunnere Livsstil Hos Innvandrer Kvinner (ASLI)
Brief Title: Empowering Immigrant Women for Active and Healthy Lifestyle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Collaborators: Oslo Municipality (Other Government); Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Ahmed A. Madar, Researcher, University of Oslo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 724880 NSD; 296558/H40 (Other: Research Council of Norway)
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Body Weight Changes; Physical Activity; Blood Glucose; Cholesterol, Elevated
MeSH Terms: conditions — Body Weight Changes; Motor Activity; Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Cluster intervenrion trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): culturally tailored intervention package on changes in lifestyle-habits
  Interventions: Behavioral: Lifestyle intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle intervention — on physical activity and healthier eating
  Arms: Intervention

SUMMARY:
The study will include overweight and obese otherwise healthy women, recruited from two main borough in Oslo with the highest population of Somali origin. The study comprises two phases: A 12-months controlled trial where the participants in the intervention borough will be compared to participants in the control borough. This is followed by a 12-months maintaining phase for the intervention borough where the control group will be given the same intervention as the intervention group received during the first 12-months.

DETAILED DESCRIPTION:
Through a research-based intervention program, the overall goal of this project is to promote immigrant health by improving, evolving and adapting a preventive healthcare in the municipality. There is social inequalities and geographical differences in health in Norway. Immigrant women struggle more with overweight and obesity than ethnic Norwegian women, and immigrant women have an increased susceptibility for diabetes and other lifestyle related diseases. In this study, we will measure the effect of a culturally tailored intervention package (physical activity and nutrition) on weight reduction, and cardio-metabolic outcomes, among overweight and obese Somali women. The study will include women (aged 20-67 years) recruited from two boroughs in Oslo with the highest population of Somali origin.

The intervention program composes a 12-month controlled trial. The core component of the program is to counsel and empower women through individual counseling and group education sessions with emphasis on physical activities and the creation of an enabling environment. The goal is that the participants become more physically active, less sedentary, eat healthy, and maintain these changes long term.

All main analysis will be done at data collected at the one-year follow up. In addition, the control group in intervention phase will after the completion of the one-year follow up be given the same intervention as the intervention group.

User involvement is included in the development, planning, implementation and dissemination of the program results. The program will produce evidence, relevant for policy-makers and stakeholders locally and globally, of how to improve health and nutrition strategies towards immigrants and minorities. The program represents a collaboration between Oslo municipality, the University of Oslo and the Norwegian School of Sport Sciences.

ELIGIBILITY:
Inclusion Criteria:

* Women living in the two boroughs in Oslo with Somali background (born in Somali regions or women born in Norway by two Somali parents), aged 20-67 years
* Being overweight or obese (BMI ≥27 kg/m2)
* Not planning to move away from the recruitment area within the next 2 years
* Not physically active on a regular basis
* Willing and able to participate in all aspects of the study
* Must be capable and willing to sign written informed consent and thumb-print for illiterate participants -

Exclusion Criteria:

* Currently pregnant
* Participating in a formal exercise or weight loss programme
* Suffering from serious bone or joint problems or difficulty walking
* Having known chronic diseases such as diabetes, cancer and uncontrolled hypo- or hyperthyroidism
* Suffering from other illnesses or being on medications that may affect weight loss
* Suffering from eating disorders
* Planning to be out of town for more than 6 weeks in the next 12 months

Ages: 20 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight in kilograms | 1 year
  Difference in weight change between intervention and control group

SECONDARY OUTCOMES:
Change in sedentary time (min/day) | 1 year
  As measured by ActivePal
Change moderately intense physical activity (min/day) | 1 year
  As measured by ActivePal
Change blood pressure | 1 year
  as measured by automatic blood pressure measuring device
Change the blood concentration of HbA1c (mmol/mol) | 1 year
  measured by blood tests
Change the blood concentration of cholesterol (total, LDL and HDL) (mmol/L) | 1 year
  measured by blood tests
Change the blood concentration of triglycerides (mmol/L) | 1 year
  measured by blood tests

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Madar, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data protection legislation makes it difficult to share individual data from this study which is limited to approx. 200 participants

REFERENCES:
- [Derived] Andersen E, Bohler L, Leirbakk MJ, Cabral D, Wedegren MC, Wieland ML, Meyer HE, Madar AA. Effects of a lifestyle programme on accelerometer-measured physical activity level and sedentary time on overweight and obese women of Somali background living in Norway. BMC Public Health. 2025 Apr 7;25(1):1310. doi: 10.1186/s12889-025-22475-z. PMID 40197263
- [Derived] Bohler L, Meyer HE, Stigum H, Leirbakk MJ, Cabral D, Wedegren MC, Andersen E, Wieland ML, Madar AA. A controlled weight loss intervention study among women of Somali background in Norway. J Migr Health. 2024 May 4;9:100231. doi: 10.1016/j.jmh.2024.100231. eCollection 2024. PMID 38766513